CLINICAL TRIAL: NCT03891485
Title: Nivolumab in mRCC Patients: Treg Function, T-cell Access and NK Interactions to Predict and Improve Efficacy
Acronym: REVOLUTION
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: 21/16 oss
Record Dates: First submitted 2019-02-26; First posted 2019-03-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-03

CONDITIONS: RCC; Metastatic Renal Cell Carcinoma
Keywords: Nivolumab; CXCR4 antagonist; mRCC; Tregs-NKs
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Archival FFPE specimen.
  Blood samples performed during standard visits and not requiring additional blood tests:
  * Heparin blood
  * EDTA blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Immunological and tumour characterization — FFPE, blood samples (liquid biopsy, heparin and EDTA blood) performed in patients presenting a renal metastatic cancer receiving treatment as standard practice according to physician's choice (2nd or 3rd line of treatment with nivolumab, or other second line according to physician's choice)

SUMMARY:
The project aims to identify Nivolumab predictive biomarkers in metastatic renal cancer patients through functional evaluation of peripheral Tregs and NKs. Moreover the efficacy of new CXCR4 antagonists (PCT/IB2011/000120/ EP2528936B1/ US2013/0079292A1) will be ex vivo evaluated in modulating Tregs and NKs function

DETAILED DESCRIPTION:
Renal cell carcinomas (RCCs) is a disease with an estimated 338,000 new cases diagnosed worldwide. Approximately 30% of patients present with metastatic disease. Since November 2015 the human IgG4 anti-PD-1 monoclonal antibody, Nivolumab, was approved to treat advanced (metastatic) clear cell renal cell carcinoma (ccRCC) patients who have received a prior anti-angiogenic therapy. PD-1 (also know as CD279), is an immune checkpoint receptor (ICR) expressed on the surface of T cells. The binding with its ligands PD-L1 (B7-H1) and PD-L2 (B7-DC) expressed on tumour cells, stromal cells or both suppress effector T cells activation and inflammatory activity promoting self-tolerance and allowing cancer cells to evade immune system. Despite encouraging results in multiple solid tumors the clinical anti-PD1 response is not as wide as expected due to multiple immuno-escape mechanisms; moreover there aren't biomarkers to predict or follow RCC patient's response to Nivolumab.

Immune evasion comprise the recruitment of immunosuppressive cells and reduced access of T-effector cells to tumor microenvironment. T-regulatory cells (Tregs) suppress a whole range of immune cells and ICRs regulate generation and/or suppression of their function. Immune cell access to tumor is controlled by the chemokine CXCL12, CXCR4 ligand. CXCL12 repels tumor-specific effector T cells and recruits suppressive cell populations at tumor sites. von Hippel-Lindau (VHL) gene mutations, detectable in 70% of RCC patients, regulate immune response inducing PD-L1 expression and promoting Natural Killer (NK) cells function. Thus NK function is a crucial element in nivolumab sensitivity.

The project will enroll patients receiving Nivolumab in 2nd or 3rd line treatment for metastatic ccRCC and, as control cohorts, either everolimus or axitinib.

Aims of the project are:

* To evaluate Tregs function on peripheral blood/neoplastic tissue from mRCC patients undergoing nivolumab treatment. Ex vivo effect of CXCR4 antagonists (PCT/IB2011/000120/ EP2528936B1/ US2013/0079292A1) and other Tregs targets antagonists (ICOS,CD39/CD73) or agonists (TLR7L) as putative anti-PD1 resistance mechanisms
* To evaluate NK function on peripheral blood/neoplastic tissue from mRCC patients undergoing nivolumab treatment. Ex vivo effect of CXCR4 antagonists

ELIGIBILITY:
Men and women with histological confirmation of advanced/metastatic RCC with not more than 2 previous therapy lines

Inclusion Criteria:

* Age ≥ 18 years-old.
* Histology proven locally advanced (unresectable) or metastatic clear cell renal cell carcinoma (mccRCC).
* Starting 2nd or 3rd line of treatment with nivolumab, everolimus or axitinib
* Signed informed consent.

Exclusion Criteria:

* Psychological, familial, sociological, geographical conditions that would limit compliance with study protocol requirements.
* Pregnant or breastfeeding woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women with histological confirmation of advanced/metastatic RCC
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Tregs function on peripheral blood/neoplastic tissue from mRCC patients undergoing nivolumab treatment. | Evolution between inclusion up to 24 months
  Treg function will be mesured as % inhibition of T-effector proliferation (Tregs/T-effector 1:1 ratio). %T-effector proliferation in the presence of patients derived Tregs (Tregs/T-effector 1:1). Ex vivo effect of CXCR4 antagonists ( PCT/IB2011/000120; EP 2 528 936 B1/US2013/0079292A1) and other Tregs targets antagonists (ICOS, CD39/CD73) or agonists (TLR7L) will be assessed to identify novel anti-PD1 resistance mechanisms.
NK function/cytotoxicity on peripheral blood/neoplastic tissue from mRCC patients undergoing nivolumab treatment | Evolution between inclusion and up to 24 months
  NK cytotoxicity will be measured as % NK cell degranulation (CD107a assay), intracellular staining Grz A and GrzB and intracellular cytokines, GM-CSF, IFNγ, IL-10, TNF. Ex vivo effect of CXCR4 antagonists will be evaluated on NK cytotoxicity.

SECONDARY OUTCOMES:
Exploration of the biological rationale for coupling CXCR4 antagonist with anti-PD-1 in in vivo models of RCC (mice models) | 36 months
  The effect of anti-PD1 and CXCR4 antagonists on tumor and tumor microenvironment cells will be evaluated in:
  * Immunocompetent model (RENCA): % tumor growth; % positive cells Granzyme/ Foxp3
  * Human xenograft model (786 cell): % tumor growth

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Nazionale Tumori di Napoli, Naples, Italy